CLINICAL TRIAL: NCT01796756
Title: Quality Improvement in Handover of General Internal Medicine In-patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Medical Protective Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H11-03542
Record Dates: First submitted 2013-02-14; First posted 2013-02-22 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Quality Improvement in Patient Handoff
Keywords: Handover; Handoff; Signout; Quality Improvement; General Internal Medicine

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Handover program (Experimental): Standardized handover program Dedicated place and time Template Face-to-face communication Evidence-based education session Feedback and audit
  Interventions: Other: Handover program
- Usual handover practice (No Intervention)

INTERVENTIONS:
Other: Handover program
  Arms: Handover program

SUMMARY:
Miscommunication during patient handover can jeopardize patient safety and is the focus of Quality Improvement initiatives by many organizations. It is widely recognized that such miscommunication is preventable using a number of strategies identified in the literature.

Currently, there is no formal handover process of General Internal Medicine in-patients, otherwise known as the Clinical Teaching Unit (CTU) at Vancouver General Hospital, which is a major patient safety concern. This project will implement a formal handover program and evaluate whether there are changes in resident satisfaction with handover, but more importantly, whether the investigators can improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Residents, medical students, and patients
* Residents and medical students will be any rotating through General Internal Medicine at Vancouver General Hospital
* Patients will be any admitted to General Internal Medicine and cared for during on-call hours (defined as 18:00 - 07:00)

Exclusion Criteria:

* None for residents and medical students
* Patients who are not being cared for during on-call hours (defined as 18:00 - 07:00)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1168 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients handed over to the on-call resident/Clinical Associate (CA) | 5 months

OTHER OUTCOMES:
Proportion of patients the resident on-call did not receive information on that would have been useful | 5 months
Frequency of patients transferred to the ICU | 5 months
Frequency of patients referred to the Critical Care Outreach Team | 5 months
Frequency of inappropriate code blue calls for patients with a "do not resuscitate" order | 5 months
Aggregate length of stay of patients admitted to the Clinical Teaching Unit | 5 months
Aggregate rate of death of patients admitted to the Clinical Teaching Unit | 5 months
Resource Utilization for patients assessed by the resident on-call overnight | 5 months
  Resource utilization will be defined by the ordering of: radiological imaging, blood work, electrocardiogram, blood transfusions, IV fluid administration, and antibiotics.

CONTACTS AND LOCATIONS:
Overall Officials: Penny Tam, BSc, MD, Principal Investigator — Vancouver General Hospital
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Tam P, Nijjar AP, Fok M, Little C, Shingina A, Bittman J, Raghavan R, Khan NA. Structured patient handoff on an internal medicine ward: A cluster randomized control trial. PLoS One. 2018 Apr 19;13(4):e0195216. doi: 10.1371/journal.pone.0195216. eCollection 2018. PMID 29672526